CLINICAL TRIAL: NCT03031782
Title: A Three-part Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Secukinumab Treatment in Juvenile Idiopathic Arthritis Subtypes of Psoriatic and Enthesitis-related Arthritis
Brief Title: Secukinumab Safety and Efficacy in Juvenile Psoriatic Arthritis (JPsA) and Enthesitis-related Arthritis (ERA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2304; 2016-003761-26 (EudraCT Number)
Record Dates: First submitted 2016-11-02; First posted 2017-01-26 (Estimated); Results first posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Juvenile Psoriatic Arthritis; Enthesitis-related Arthritis
Keywords: JIA; JPsA; ERA; Secukinumab; ILAR; Arthritis
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Period 2 - active (Experimental): secukinumab (AIN457 - pre-filled syringe) for patients with a minimum American college of Rheumatology (ACR) 30 response in Treatment Period 1
  Interventions: Drug: secukinumab
- Treatment Period 2 - placebo (Placebo Comparator): placebo comparator (matched to secukinumab treatment) for patients with a minimum American college of Rheumatology (ACR) 30 response in Treatment Period 1
  Interventions: Other: placebo

INTERVENTIONS:
Drug: secukinumab — secukinumab is a high-affinity fully human monoclonal anti-human antibody that targets IL-17A and neutralizes activity.
  Other Names: AIN457
  Arms: Treatment Period 2 - active
Other: placebo — Matched placebo to AIN457 for use in the double blind Treatment Period 2
  Arms: Treatment Period 2 - placebo

SUMMARY:
This was a double-blind, placebo-controlled, event-driven randomized withdrawal study to investigate the efficacy and safety of secukinumab treatment in the Juvenile Idiopathic Arthritis (JIA) categories of Juvenile Psoriatic Arthritis (JPsA) and Enthesitis-related Arthritis (ERA). The study was divided into 3 parts (plus a post-treatment follow-up period) consisting of open-label, single-arm active treatment in Treatment Periods 1 and 3 and a randomized, double-blind, placebo controlled, event-driven withdrawal design in Treatment Period 2

DETAILED DESCRIPTION:
TP1: All eligible subjects entered TP1 to receive 12-weeks of open-label secukinumab at a dose predicted to achieve secukinumab serum levels equivalent to adults administered a 150 mg dose regimen. Secukinumab was administered s.c. weekly for the first 4 weeks (Baseline, Weeks 1, 2, 3, 4) and then every 4 weeks thereafter. Clinical response (JIA ACR 30) was assessed at Week 12. Responders advanced to TP2 and non-responders exited the trial (early termination visit and entered into the Post-treatment follow-up period).

TP2: Subjects who were a responder (JIA ACR 30) at Week 12 entered the double-blind withdrawal TP2 and were randomized 1:1 to either secukinumab or placebo on that visit and then every 4 weeks, until either experiencing a disease flare or completion of TP2. TP2 was event driven and was planned to be closed when 33 subjects experienced a disease flare as per JIA definition. Alternatively, the study could be closed when all subjects reached the total study duration of 104 Weeks and therefore subjects who did not experience a disease flare remained in TP2 for the duration of the study and completed the study without entering into TP3

TP3: Subjects experiencing a disease flare in TP2 immediately entered TP3 to receive openlabel secukinumab every 4 weeks until total study duration of 104 weeks for that subject was achieved.

Post-treatment follow-up: The post-treatment follow-up period (lasting 12 weeks from the last study drug administration) was required for all subjects, unless they qualified and entered the secukinumab extension trial. All subjects were expected to participate in the post-treatment follow up period, except for those entering the extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Enthesitis-related arthritis (ERA) or Juvenile psoriatic arthritis (JPsA) according to the International League of Associations for Rheumatology (ILAR) classification criteria of at least 6 months duration.
2. Active disease (ERA or JPsA) defined as having both:

   * at least 3 active joints
   * at least 1 site of active enthesitis at baseline or documented by history.
3. Inadequate response (at least 1 month) or intolerance to at least 1 nonsteroidal anti-inflammatory drugs(NSAID)
4. Inadequate response (at least 2 months) or intolerance to at least 1 Disease-modifying antirheumatic drugs (DMARD)
5. No concomitant use of second line agents such as disease-modifying and/or immunosuppressive drugs.

Exclusion Criteria:

1. Patients fulfilling any ILAR diagnostic JIA category other than ERA or JPsA.
2. Patients who have ever received biologic immunomodulating agents
3. Patients taking any non-biologic DMARD except for MTX (or sulfasalazine for ERA patients only).
4. Patients with active uncontrolled inflammatory bowel disease or active uncontrolled uveitis.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (4):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Portland, Oregon
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Laken
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Saint Augustin
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Krakow, Poland
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yekaterinburg
- South Africa (2):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Panorama
- Spain (2):
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Valencia
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, Halkali
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
- United Kingdom (5):
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Weiss PF, Ruperto N, Quebe-Fehling E, Shew A, Pricop L, Pieterse CC, Brunner HI; Paediatric Rheumatology International Trials Organisation (PRINTO) and Pediatric Rheumatology Collaborative Study Group (PRCSG) Investigative Sites. Juvenile Spondyloarthritis Disease Activity Index Validation in Enthesitis-Related Arthritis and Juvenile Psoriatic Arthritis in a Prospective Clinical Trial Setting. J Rheumatol. 2026 Jan 1;53(1):85-94. doi: 10.3899/jrheum.2025-0294. PMID 40953957
- [Derived] Brunner HI, Foeldvari I, Alexeeva E, Ayaz NA, Calvo Penades I, Kasapcopur O, Chasnyk VG, Hufnagel M, Zuber Z, Schulert G, Ozen S, Rakhimyanova A, Ramanan A, Scott C, Sozeri B, Zholobova E, Martin R, Zhu X, Whelan S, Pricop L, Martini A, Lovell D, Ruperto N; Paediatric Rheumatology INternational Trials Organization (PRINTO) and Pediatric Rheumatology Collaborative Study Group (PRCSG). Secukinumab in enthesitis-related arthritis and juvenile psoriatic arthritis: a randomised, double-blind, placebo-controlled, treatment withdrawal, phase 3 trial. Ann Rheum Dis. 2023 Jan;82(1):154-160. doi: 10.1136/ard-2022-222849. Epub 2022 Aug 12. PMID 35961761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 86 subjects entered TP1
Pre-assignment Details: AIN457 treatment group refers to all subjects who did not take any placebo before or during the period in the study. The term Placebo in TP2 refers to all subjects who took placebo in TP2 and secukinumab in other periods. For ease of reading, Placebo in TP2 treatment group is referred as placebo treatment group or placebo hereafter in this document.
Groups:
- AIN457 in TP1: Treatment Period 1
- AIN457 in TP 2: Treatment Period 2
- Placebo in TP2: Includes all participants who received placebo, i.e. were randomized to Placebo in TP2. In this arm, AEs are reported for all three treatment periods (TP1, TP2 and TP3) combined, i.e. also including AEs that occurred when treated with AIN457 in TP1 or TP3.
- AIN457 in TP3; Placebo in TP 3: Treatment Period 3
Period: Treatment Period 1
Arm/Group | AIN457 in TP1 | AIN457 in TP 2 | Placebo in TP2 | AIN457 in TP3 | Placebo in TP 3
Started | 86 | 0 | 0 | 0 | 0
Completed | 83 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | AIN457 in TP1 | AIN457 in TP 2 | Placebo in TP2 | AIN457 in TP3 | Placebo in TP 3
Started | 0 | 37 | 38 | 0 | 21
Completed | 0 | 31 | 36 | 0 | 16
Not Completed | 0 | 6 | 2 | 0 | 5
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0
Period: Treatment Period 3
Arm/Group | AIN457 in TP1 | AIN457 in TP 2 | Placebo in TP2 | AIN457 in TP3 | Placebo in TP 3
Started | 0 | 0 | 0 | 11 | 0
Completed | 0 | 0 | 0 | 10 | 0
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included subjects who received any treatment. TP1 = 86, TP2 = 75
Groups:
- All Participants: TP1 open-label: Secukinumab 75 mg or 150 mg based on the body weight (<50 kg or >= 50 kg) was administered s.c. At Week 12 (end of TP1), subject's response to study drug was determined (responders entered TP2 and non-responders entered post-treatment follow-up)
Arm/Group | All Participants
Number analyzed (Participants) | 86
Age, Categorical [Count of Participants; unit: Participants] — Population: Safety Set
  Participants
    AIN457 in Treatment Period 1: <=18 years | 86
    AIN457 in Treatment Period 1: Between 18 and 65 years | 0
    AIN457 in Treatment Period 1: >=65 years | 0
    AIN457 in Treatment Period 2: number analyzed (Participants) | 37
    AIN457 in Treatment Period 2: <=18 years | 37
    AIN457 in Treatment Period 2: Between 18 and 65 years | 0
    AIN457 in Treatment Period 2: >=65 years | 0
    placebo in TP2: number analyzed (Participants) | 38
    placebo in TP2: <=18 years | 38
    placebo in TP2: Between 18 and 65 years | 0
    placebo in TP2: >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age of participants in years
  ERA + JPsA = Total Population: Safety Set
  years
    AIN457 in Treatment Period 1 - JIA Category: ERA: number analyzed (Participants) | 52
    AIN457 in Treatment Period 1 - JIA Category: ERA | 13.7 (2.62)
    AIN457 in Treatment Period 1 - JIA Category: JPsA: number analyzed (Participants) | 34
    AIN457 in Treatment Period 1 - JIA Category: JPsA | 12.2 (3.66)
    AIN457 in Treatment Period 2 - JIA Category: ERA: number analyzed (Participants) | 22
    AIN457 in Treatment Period 2 - JIA Category: ERA | 14 (2.46)
    AIN457 in Treatment Period 2 - JIA Category: JPsA: number analyzed (Participants) | 16
    AIN457 in Treatment Period 2 - JIA Category: JPsA | 13.1 (3.14)
    Placebo in TP2- JIA Category: ERA: number analyzed (Participants) | 22
    Placebo in TP2- JIA Category: ERA | 13 (2.94)
    Placebo in TP2 - JIA Category JPsA: number analyzed (Participants) | 16
    Placebo in TP2 - JIA Category JPsA | 10.6 (3.70)
Sex: Female, Male [Count of Participants; unit: Participants] — ERA + JPsA = Total Population: Safety Set
  Participants
    AIN457 in Treatment Period 1 - JIA Category: ERA: number analyzed (Participants) | 52
    AIN457 in Treatment Period 1 - JIA Category: ERA: Female | 11
    AIN457 in Treatment Period 1 - JIA Category: ERA: Male | 41
    AIN457 in Treatment Period 1 -JIA Category: JPsA: number analyzed (Participants) | 34
    AIN457 in Treatment Period 1 -JIA Category: JPsA: Female | 18
    AIN457 in Treatment Period 1 -JIA Category: JPsA: Male | 16
    AIN457 in Treatment Period 2 - JIA Category: ERA: number analyzed (Participants) | 22
    AIN457 in Treatment Period 2 - JIA Category: ERA: Female | 4
    AIN457 in Treatment Period 2 - JIA Category: ERA: Male | 18
    AIN457 in Treatment Period 2 -JIA Category: JPsA: number analyzed (Participants) | 15
    AIN457 in Treatment Period 2 -JIA Category: JPsA: Female | 9
    AIN457 in Treatment Period 2 -JIA Category: JPsA: Male | 6
    Placebo in TP2 - JIA Category: ERA: number analyzed (Participants) | 22
    Placebo in TP2 - JIA Category: ERA: Female | 4
    Placebo in TP2 - JIA Category: ERA: Male | 18
    Placebo in TP2 - JIA Category: JPsA: number analyzed (Participants) | 16
    Placebo in TP2 - JIA Category: JPsA: Female | 7
    Placebo in TP2 - JIA Category: JPsA: Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — ERA + JPsA = Total
  Unknown or Not Reported Row also means "Other" (none of the above) Population: Safety Set
  Participants
    AIN457 in Treatment Period 1 - JIA Category: ERA: number analyzed (Participants) | 52
    AIN457 in Treatment Period 1 - JIA Category: ERA: American Indian or Alaska Native | 0
    AIN457 in Treatment Period 1 - JIA Category: ERA: Asian | 0
    AIN457 in Treatment Period 1 - JIA Category: ERA: Native Hawaiian or Other Pacific Islander | 0
    AIN457 in Treatment Period 1 - JIA Category: ERA: Black or African American | 0
    AIN457 in Treatment Period 1 - JIA Category: ERA: White | 51
    AIN457 in Treatment Period 1 - JIA Category: ERA: More than one race | 0
    AIN457 in Treatment Period 1 - JIA Category: ERA: Unknown or Not Reported | 1
    AIN457 in Treatment Period 1 - JIA Category: JPsA: number analyzed (Participants) | 34
    AIN457 in Treatment Period 1 - JIA Category: JPsA: American Indian or Alaska Native | 0
    AIN457 in Treatment Period 1 - JIA Category: JPsA: Asian | 1
    AIN457 in Treatment Period 1 - JIA Category: JPsA: Native Hawaiian or Other Pacific Islander | 0
    AIN457 in Treatment Period 1 - JIA Category: JPsA: Black or African American | 0
    AIN457 in Treatment Period 1 - JIA Category: JPsA: White | 31
    AIN457 in Treatment Period 1 - JIA Category: JPsA: More than one race | 0
    AIN457 in Treatment Period 1 - JIA Category: JPsA: Unknown or Not Reported | 2
    AIN457 in Treatment Period 2 - JIA Category: ERA: number analyzed (Participants) | 22
    AIN457 in Treatment Period 2 - JIA Category: ERA: American Indian or Alaska Native | 0
    AIN457 in Treatment Period 2 - JIA Category: ERA: Asian | 0
    AIN457 in Treatment Period 2 - JIA Category: ERA: Native Hawaiian or Other Pacific Islander | 0
    AIN457 in Treatment Period 2 - JIA Category: ERA: Black or African American | 0
    AIN457 in Treatment Period 2 - JIA Category: ERA: White | 22
    AIN457 in Treatment Period 2 - JIA Category: ERA: More than one race | 0
    AIN457 in Treatment Period 2 - JIA Category: ERA: Unknown or Not Reported | 0
    AIN457 in Treatment Period 2 - JIA Category: JPsA: number analyzed (Participants) | 15
    AIN457 in Treatment Period 2 - JIA Category: JPsA: American Indian or Alaska Native | 0
    AIN457 in Treatment Period 2 - JIA Category: JPsA: Asian | 0
    AIN457 in Treatment Period 2 - JIA Category: JPsA: Native Hawaiian or Other Pacific Islander | 0
    AIN457 in Treatment Period 2 - JIA Category: JPsA: Black or African American | 14
    AIN457 in Treatment Period 2 - JIA Category: JPsA: White | 0
    AIN457 in Treatment Period 2 - JIA Category: JPsA: More than one race | 0
    AIN457 in Treatment Period 2 - JIA Category: JPsA: Unknown or Not Reported | 1
    Placebo in TP2 - JIA Category: ERA: number analyzed (Participants) | 22
    Placebo in TP2 - JIA Category: ERA: American Indian or Alaska Native | 0
    Placebo in TP2 - JIA Category: ERA: Asian | 0
    Placebo in TP2 - JIA Category: ERA: Native Hawaiian or Other Pacific Islander | 0
    Placebo in TP2 - JIA Category: ERA: Black or African American | 0
    Placebo in TP2 - JIA Category: ERA: White | 21
    Placebo in TP2 - JIA Category: ERA: More than one race | 0
    Placebo in TP2 - JIA Category: ERA: Unknown or Not Reported | 1
    Placebo in TP2 - JIA Category: JPsA: number analyzed (Participants) | 16
    Placebo in TP2 - JIA Category: JPsA: American Indian or Alaska Native | 0
    Placebo in TP2 - JIA Category: JPsA: Asian | 0
    Placebo in TP2 - JIA Category: JPsA: Native Hawaiian or Other Pacific Islander | 1
    Placebo in TP2 - JIA Category: JPsA: Black or African American | 0
    Placebo in TP2 - JIA Category: JPsA: White | 14
    Placebo in TP2 - JIA Category: JPsA: More than one race | 0
    Placebo in TP2 - JIA Category: JPsA: Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Flare During Treatment Period 2
Description: Survival analysis of time to flare in treatment period 2 (TP2) FAS2
  Subjects are either ERA or JPsA
Time Frame: From Week 12 until max Week 104
Population: Full Analysis Set for TP2: The FAS TP2 (FAS 2) consisted of all randomized subjects who received at least one dose of study drug in TP2. Following the intent-to-treat principle, subjects were analyzed according to the treatment they were assigned to at randomization in TP2.
Measure: Count of Participants; unit: Participants
Groups:
- AIN457 in Treatment Period 2: Includes all participants who did not receive placebo, i.e. either did not enter TP2 or were randomized to AIN457 in TP2. In this arm, AEs are reported for all three treatment periods (TP1, TP2 and TP3) combined.
Arm/Group | AIN457 in Treatment Period 2 | Placebo in TP2
Number analyzed (Participants) | 37 | 38
Participants | 10 | 21
Statistical Analysis 1: Comparison: AIN457 in Treatment Period 2 vs Placebo in TP2; Survival analysis of time to flare - TP2 (FAS2); Test type: Superiority; p < 0.001, Log Rank; Hazard ratios and associated 95% confidence intervals are based on a Cox proportional hazards model with treatment and analysis factors; Cox Proportional Hazard = 0.28, 95% CI 2-sided [0.13 to 0.63]

2. Secondary Outcome: Percent of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30/50/70/90/100 Response at Week 12 - by JIA Category
Description: Summary of JIA ACR 30/50/70/90/100 for all subjects and each JIA category - TP1 (FAS1)
  The adapted ACR Pediatric 30/50/70/90/100 criteria was used to determine efficacy defined as improvement from baseline of at least 30/50/70/90/100% respectively in at least 3 of the following 6 components
  * Physician's Global Assessment of disease activity on a 0-100 mm VAS from 0 mm = no disease activity to 100 mm = very severe disease activity.
  * Parent's or patient's Global Assessment of Subject's overall wellbeing on a 0-100 mm VAS from 0 mm= very well to 100 mm= very poor.
  * Functional ability: Childhood Health Assessment Questionnaire (CHAQ©)
  * Number of joints with active arthritis using the ACR definition (The ACR definition of active arthritis is any joint with swelling, or in the absence of swelling, limitation of motion accompanied by either pain on motion or tenderness not due to deformity)
  * Number of joints with limitation of motion
  * Laboratory measure of inflammation: CRP (mg/L)
Time Frame: baseline, week 12
Population: Full Analysis Set for TP1: The FAS TP1 (FAS 1) consisted of all subjects who received at least one dose of study drug in TP1.
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- AIN457 in Treatment Period 1 - ERA: TP1 open-label: Secukinumab 75 mg or 150 mg based on the body weight (<50 kg or >= 50 kg) was administered s.c. end of TP1 visit at week 12 was determined based on subject's response to the study drug administered (responders entered TP2 and non-responders entered post-treatment follow-up)
- AIN457 in Treatment Periiod 1 - JPsA: TP1 open-label: Secukinumab 75 mg or 150 mg based on the body weight (<50 kg or >+ 50 kg) was administered s.c. end of TP1 visit at week 12 was determined based on subject's response to the study drug administered (responders entered TP2 and non-responders entered post-treatment follow-up)
Arm/Group | AIN457 in Treatment Period 1 - ERA | AIN457 in Treatment Periiod 1 - JPsA
Number analyzed (Participants) | 52 | 34
percent of participants
  ACR 30: number analyzed (Participants) | 51 | 32
  ACR 30 | 86.3 [73.1 to 93.8] | 96.9 [82.0 to 99.8]
  ACR 50: number analyzed (Participants) | 51 | 32
  ACR 50 | 80.4 [66.5 to 89.7] | 96.9 [82.0 to 99.8]
  ACR 70: number analyzed (Participants) | 51 | 32
  ACR 70 | 66.7 [52.0 to 78.9] | 75.0 [56.2 to 87.9]
  ACR 90: number analyzed (Participants) | 51 | 32
  ACR 90 | 33.3 [21.1 to 48.0] | 50.0 [32.2 to 67.8]
  ACR 100: number analyzed (Participants) | 51 | 32
  ACR 100 | 27.5 [16.3 to 42.0] | 21.9 [9.9 to 40.4]

3. Secondary Outcome: Percent of Participants With Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30/50/70/90/100 Response at Week 12 - Total
Description: Summary of JIA ACR 30/50/70/90/100 for all subjects - TP1 (FAS1)
  The adapted ACR Pediatric 30/50/70/90/100 criteria was used to determine efficacy defined as improvement from baseline of at least 30/50/70/90/100% respectively in at least 3 of the following 6 components
  * Physician's Global Assessment of disease activity on a 0-100 mm VAS from 0 mm = no disease activity to 100 mm = very severe disease activity.
  * Parent's or patient's Global Assessment of Subject's overall wellbeing on a 0-100 mm VAS from 0 mm= very well to 100 mm= very poor.
  * Functional ability: Childhood Health Assessment Questionnaire (CHAQ©)
  * Number of joints with active arthritis using the ACR definition (The ACR definition of active arthritis is any joint with swelling, or in the absence of swelling, limitation of motion accompanied by either pain on motion or tenderness not due to deformity)
  * Number of joints with limitation of motion
  * Laboratory measure of inflammation: CRP (mg/L)
Time Frame: baseline, week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- AIN457 in Treatment Period 1 - TOTAL: TP1 open-label: Secukinumab 75 mg or 150 mg based on the body weight (<50 kg or >= 50 kg) was administered s.c. end of TP1 visit at week 12 was determined based on subject's response to the study drug administered (responders entered TP2 and non-responders entered post-treatment follow-up)
Arm/Group | AIN457 in Treatment Period 1 - TOTAL
Number analyzed (Participants) | 86
percent of participants
  ACR 30: number analyzed (Participants) | 83
  ACR 30 | 90.4 [81.4 to 95.4]
  ACR 50: number analyzed (Participants) | 83
  ACR 50 | 86.7 [77.1 to 92.9]
  ACR 70: number analyzed (Participants) | 51
  ACR 70 | 69.9 [58.7 to 79.2]
  ACR 90: number analyzed (Participants) | 51
  ACR 90 | 39.8 [29.4 to 51.1]
  ACR 100: number analyzed (Participants) | 51
  ACR 100 | 25.3 [16.7 to 36.2]

4. Secondary Outcome: Percent Change From Baseline for JIA ACR Core Components in TP1
Description: Summary of JIA ACR core components for all subjects and each JIA category - Treatment period 1
  Negative percent change indicates improvement
  Physician global assessment of disease activity (VAS mm) 0 (no disease activity) - 100 (very severe); Parent or subject global assessment of overall well-being (VAS mm) 0 (very well) - 100 (very poor); CHAQ (Childhood Health Assessment Questionnaire) 0 - 3 (most severe); Number of joints with active arthritis 0 - 73; Number of joints with limited range of motion 0 - 69.
Time Frame: baseline, week 12
Population: FAS TP1 including patients with valid measurements at week 12
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- AIN457 in Treatment Period 1: TP1 open-label: Secukinumab 75 mg or 150 mg based on the body weight (<50 kg or >= 50 kg) was administered s.c. end of TP1 visit at week 12 was determined based on subject's response to the study drug administered (responders entered TP2 and non-responders entered post-treatment follow-up)
Arm/Group | AIN457 in Treatment Period 1
Number analyzed (Participants) | 86
percent change
  physician global assessment of disease activity: number analyzed (Participants) | 83
  physician global assessment of disease activity | -77.4 (22.67)
  parent/subject global assessment of overall well-being: number analyzed (Participants) | 83
  parent/subject global assessment of overall well-being | -53.1 (58.43)
  functional ability (CHAQ): number analyzed (Participants) | 83
  functional ability (CHAQ) | -53.776 (70.5034)
  number of joints with active arthritis: number analyzed (Participants) | 83
  number of joints with active arthritis | -79.3 (34.86)
  number of joints with limited range of motion: number analyzed (Participants) | 83
  number of joints with limited range of motion | -72.5 (38.19)

5. Secondary Outcome: Percent Change in C-reactive Protein Standardized Value (mg/L)
Description: Median Percent Change from baseline for C-reactive protein standardized value (mg/L)
Time Frame: baseline, week 12
Population: FAS TP1
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | AIN457 in Treatment Period 1
Number analyzed (Participants) | 82
percent change | -13.587 (227.6901)

6. Secondary Outcome: Change From Baseline Juvenile Arthritis Disease Activity Score (JADAS) Score
Description: JADAS change from baseline for all subjects in Treatment period 1. JADAS-27 (Juvenile Arthritis Disease Activity Score in 27 joints) ranges from 0 to 57 and JADAS-71 ranges from 0 to 101 (higher scores indicate more disease activity).
Time Frame: 12 weeks
Population: FAS treatment period 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | AIN457 in Treatment Period 1
Number analyzed (Participants) | 86
score
  JADAS-27: number analyzed (Participants) | 83
  JADAS-27 | -10.487 (7.2262)
  JADAS-71: number analyzed (Participants) | 83
  JADAS-71 | -13.403 (9.7300)

7. Secondary Outcome: Change From Baseline in Total Enthesitis Events - TP1 (FAS1)
Description: Enthesitis swollen joint count range is 0-16. Zero is worst, and 16 is best
  A total of 16 entheseal sites were assessed for the presence or absence of tenderness of enthesitis.
  This is the mean (SD) enthesitis count (range 0-16) for FAS subjects
  A zero score means no enthesitis, so a zero score is better for the patient
Time Frame: Baseline and week 12
Population: FAS TP1 including patients with valid measurements at week 12
Measure: Mean (Standard Deviation); unit: Number of enthesitis events
Arm/Group | AIN457 in Treatment Period 1
Number analyzed (Participants) | 83
Number of enthesitis events | -1.8 (2.31)

8. Secondary Outcome: Change From Baseline in Total Dactylitis Count
Description: Summary of total dactylitis count for all subjects - TP1 (FAS1)
  Total dactylitis count ranges from 0 to 20. A zero score means no dactylitis, so a zero score is better for the patient
Time Frame: baseline, week 12
Population: FAS TP1 including patients with valid measurements at week 12
Measure: Mean (Standard Deviation); unit: Number of dactylitis events
Arm/Group | AIN457 in Treatment Period 1
Number analyzed (Participants) | 78
Number of dactylitis events | -0.8 (1.83)

9. Secondary Outcome: Number of Participants With Anti-secukinumab Anitbodies
Description: Blood samples for immunogenicity (anti-AIN457 antibodies) were taken pre-dose at the scheduled time points. In addition, if a subject discontinued from the study at any time, he/she provided a sample at the last visit. All blood samples were taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. An Electrochemiluminescence method was used for the detection of potential anti-secukinumab antibody formation.
Time Frame: 104 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Groups:
- AIN457 in Treatment Period 2 - Active: TP2 treatment withdrawal: Secukinumab (AIN457 - pre-filled syringe) for patients with a minimum American college of Rheumatology (ACR) 30 response in Treatment Period 1
- Placebo TP2: Placebo s.c. in Treatment Period 2: all subjects who took placebo in TP2 and AIN457 in other period/s
Arm/Group | AIN457 in Treatment Period 1 | AIN457 in Treatment Period 2 - Active | Placebo TP2
Number analyzed (Participants) | 86 | 37 | 38
Participants | 0 | 0 | 0

10. Secondary Outcome: Secukinumab Serum Concentration
Description: Summary of pharmacokinetic concentrations - Treatment period 1
Time Frame: baseline, week 12
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- AIN457 in Treatment Period 1: to week 12
  TP1 open-label: Secukinumab 75 mg or 150 mg based on the body weight (<50 kg or >= 50 kg) was administered s.c. end of TP1 visit at week 12 was determined based on subject's response to the study drug administered (responders entered TP2 and non-responders entered post-treatment follow-up)
Arm/Group | AIN457 in Treatment Period 1
Number analyzed (Participants) | 86
mcg/mL
  <50 kg | 30.9 (12.9)
  >=50 kg | 34.6 (11.2)

11. Secondary Outcome: Number of Participants With Inactive Disease Status for All Subjects - TP1 (FAS1)
Description: Summary of inactive disease status for all subjects - TP1 (FAS1)
  Clinical inactive disease definition was adapted from the JIA ACR criteria.
  All were required to be met:
  * No joints with active arthritis
  * No uveitis
  * CRP value within normal limits for the laboratory where tested or, if elevated, not attributable to JIA
  * Physician's global assessment of disease activity score ≤ 10mm
  * Duration of morning stiffness attributable to JIA ≤15 min
Time Frame: week 12
Population: FAS1
Measure: Number (95% Confidence Interval); unit: partcipants
Arm/Group | AIN457 in Treatment Period 1
Number analyzed (Participants) | 83
partcipants | 30 [26.1 to 47.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time patient provided informed consent until the end of study. Serious Adverse Events (SAEs) were collected after the patient provided informed consent and until 12 weeks after last administered dose of study treatment or 30 days after the subject has stopped study participation (whichever is later)
Description: AEs are any untoward sign or symptom that occurred during the study treatment period.
  AEs are presented across all three treatment periods combined since due to the study design, the exposure times for Placebo (only received in TP2) and Secukinumab were different over the entire treatment period. In addition, it cannot be ruled-out that events occurring in TP2 under placebo are due to a spill-over effect by the previous secukinumab treatment in TP1
Groups:
- AIN457 in Entire Treatment Period: Includes all participants who did not receive placebo, i.e. either did not enter TP2 or were randomized to AIN457 in TP2. In this arm, AEs are reported for all three treatment periods (TP1, TP2 and TP3) combined.
- Total: Includes all participants who were treated with study medication. In this arm, AEs are reported for all three treatment periods (TP1, TP2 and TP3) combined.
Arm/Group | AIN457 in Entire Treatment Period | Placebo in TP2 | Total
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/38 | 0/86
Serious Adverse Events (participants affected / at risk) | 7/48 | 4/38 | 11/86
Other Adverse Events (participants affected / at risk) | 44/48 | 35/38 | 79/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 in Entire Treatment Period (N=48) | Placebo in TP2 (N=38) | Total (N=86)
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Juvenile psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 in Entire Treatment Period (N=48) | Placebo in TP2 (N=38) | Total (N=86)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 4
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 1
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 3
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 3
Conjunctivitis allergic (Eye disorders) | 1 | 1 | 2
Eye haematoma (Eye disorders) | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1
Myopia (Eye disorders) | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 2 | 0 | 2
Uveitis (Eye disorders) | 2 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 6 | 8
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 5
Aphthous ulcer (Gastrointestinal disorders) | 4 | 1 | 5
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 11 | 6 | 17
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Lip disorder (Gastrointestinal disorders) | 1 | 0 | 1
Malpositioned teeth (Gastrointestinal disorders) | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 11 | 8 | 19
Noninfective gingivitis (Gastrointestinal disorders) | 1 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 5 | 4 | 9
Administration site reaction (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 2 | 3
Feeling hot (General disorders) | 0 | 1 | 1
Injection site erythema (General disorders) | 0 | 1 | 1
Injection site pain (General disorders) | 2 | 1 | 3
Injection site pruritus (General disorders) | 1 | 1 | 2
Injection site reaction (General disorders) | 1 | 0 | 1
Medical device pain (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 1
Peripheral swelling (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 6 | 6 | 12
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 | 1 | 2
Mite allergy (Immune system disorders) | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0 | 1
Adenoiditis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 2
Conjunctivitis (Infections and infestations) | 3 | 2 | 5
Enterobiasis (Infections and infestations) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 2 | 4
Gastrointestinal infection (Infections and infestations) | 1 | 2 | 3
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 1
Helminthic infection (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 1
Impetigo (Infections and infestations) | 1 | 3 | 4
Influenza (Infections and infestations) | 5 | 0 | 5
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Nail bed infection (Infections and infestations) | 1 | 0 | 1
Nail infection (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 16 | 11 | 27
Onychomycosis (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 2 | 3
Oral viral infection (Infections and infestations) | 0 | 1 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 1
Otitis media (Infections and infestations) | 1 | 3 | 4
Paronychia (Infections and infestations) | 3 | 1 | 4
Pharyngitis (Infections and infestations) | 6 | 3 | 9
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0 | 3
Pulpitis dental (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 4 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 2 | 2
Rhinitis (Infections and infestations) | 3 | 5 | 8
Sinusitis (Infections and infestations) | 3 | 0 | 3
Skin infection (Infections and infestations) | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 4 | 3 | 7
Tracheitis (Infections and infestations) | 2 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 10 | 9 | 19
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Vaginal infection (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 2 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 2 | 4
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 4 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Gingival injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 4 | 5
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 3 | 6
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 3 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 1 | 3
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Venomous sting (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Blood calcium increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 1 | 1
Blood pressure systolic increased (Investigations) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 1
Body temperature increased (Investigations) | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 2
Platelet count increased (Investigations) | 1 | 0 | 1
Transaminases increased (Investigations) | 1 | 2 | 3
Weight increased (Investigations) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4 | 12
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Juvenile psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 6 | 6 | 12
Nerve compression (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 1
Distractibility (Psychiatric disorders) | 0 | 1 | 1
Euphoric mood (Psychiatric disorders) | 1 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 1
Mental disorder (Psychiatric disorders) | 0 | 1 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 3 | 0 | 3
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2 | 2
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 1 | 2
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 1
Varicocele (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 12
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin striae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Sexual abuse (Social circumstances) | 1 | 0 | 1
Cyanosis (Vascular disorders) | 1 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT03031782/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT03031782/SAP_001.pdf